CLINICAL TRIAL: NCT03597412
Title: Efficacy and Safety of Rosuvastatin/Ezetimibe Combination Therapy Versus Rosuvastatin Monotherapy in Atherosclerotic Cardiovascular Disease (ASCVD) Patients With Type 2 Diabetes Mellitus (DM)
Brief Title: Rosuvastatin/Ezetimibe Versus Rosuvastatin in ASCVD Patients With Type 2 DM
Acronym: MIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC038
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Atherosclerotic Cardiovascular Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvamibe Tab (Experimental): Rosuvastatin 10mg/Ezetimibe 10mg qd for 24 weeks
  Interventions: Drug: Rosuvamibe
- Monorova Tab (Active Comparator): Rosuvastatin 20mg qd for 24 weeks
  Interventions: Drug: Monorova

INTERVENTIONS:
Drug: Rosuvamibe — Rosuvastatin 10mg/Ezetimibe 10mg
  Arms: Rosuvamibe Tab
Drug: Monorova — Rosuvastatin 20mg
  Arms: Monorova Tab

SUMMARY:
This study will evaluate the efficacy and aafety of rosuvastatin/ezetimibe combination therapy vs. rosuvastatin monotherapy in atherosclerotic cardiovascular disease patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 and above
2. Patient with type 2 diabetes taking oral diabetes medication for at least 3 months
3. Patient diagnosed with ASCVD

   * Myocardial Infarction (MI)
   * Acute coronary syndrome (ACS)
   * History of Coronary revascularization(Percutaneous Coronary Intervention, PCI)
   * History of Coronary artery bypass graft surgery (CABG) or other arterial revascularization procedures
   * Stroke or Transient ischemic attack (TIA)
   * Peripheral Arterial Disease (PAD)
   * Stable Angina
4. Written informed consent

Exclusion Criteria:

1. Type 1 diabetes
2. HbA1c > 8.5% at screening
3. Fasting triglyceride ≥ 400 mg/dL at screening
4. History of muscular disease or rhabdomyolysis due to use of statin
5. Hypersensitive to rosuvastatin or ezetemibe
6. Contraindications stated in the SPC of rosuvastatin or rosuvastatin/ezetimibe including the following:

   ① Severe renal disease (CrCL < 30mL/min: Cockcroft-gault formula or estimated GFR (MDRD) < 30mL/min/1.73m2)

   ② ALT, AST > 3x ULN or history of active liver disease

   ③ CPK > 3x ULN
7. Those participating in clinical trials of other drugs
8. Other than the above who is deemed to be ineligible to participate in the trial by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in LDL-C level | Baseline, Week 24

SECONDARY OUTCOMES:
Change from baseline to week 12 in LDL-C level | Baseline, Week 12
Change from baseline to week 12 and week 24 in total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in high-sensitivity C-reactive protein (hs-CRP) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in Apolipoprotein A1, Apolipoprotein B, Apolipoprotein B48, and Apolipoprotein B/Apolipoprotein A1 | Baseline, Week 24
Change from baseline to week 12 and week 24 in glycosylated hemoglobin (HbA1c) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in fasting plasma glucose (FPG) | Baseline, Week 12, Week 24
Change from baseline to week 12 and week 24 in homeostasis model assessment for insulin resistance (HOMA-IR) | Baseline, Week 12, Week 24
Proportion of subjects achieving LDL-C < 70mg/dL | Baseline, Week 12, Week 24
Proportion of subjects achieving LDL-C < 55mg/dL | Baseline, Week 12, Week 24
Occurrence of MACCE (Major Adverse Cardiovascular and Cerebrovascular Event) | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided